CLINICAL TRIAL: NCT02428933
Title: Dopaminergic Effects on Brown Adipose Tissue: the DEBAT Trial
Brief Title: Dopaminergic Effects on Brown Adipose Tissue
Acronym: DEBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, F Holleman, Dr. MD., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: METC nr 2013_107
Record Dates: First submitted 2014-10-17; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: Brown Adipose Tissue; Obesity; Insulin Sensitivity; Dopamine
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Before and after bromocriptine (Other): Subjects will be investigated before and after the use of bromocriptine. They will use bromocriptine for two weeks in the evening (1.25mg/day during the first week and 2.5mg/day during the second week).
  Interventions: Drug: Bromocriptine

INTERVENTIONS:
Drug: Bromocriptine — The investigators will look at the physiological effect of dopamine on BAT activity rather than on the effect of the drug itself
  Other Names: Parlodel

SUMMARY:
In this study the investigators will investigate the effect of dopamine (bromocriptine) on Brown Adipose Tissue in lean, young, healthy males.

The investigators will also examine energy expenditure, body temperature and insulin sensitivity as measurements of Brown Adipose Tissue activity.

DETAILED DESCRIPTION:
In this study the investigators will investigate whether bromocriptine influences the metabolic activity of BAT, as assessed with a 18F-fluorodeoxyglucose (18F-FDG) Positron Emission Tomography (PET)-CT scan

This is an observational, prospective design with invasive measurements. The investigators will include 16 healthy lean male volunteers (aged 18-30 years, BMI 19-25 kg/m2) The volunteers will be recruited by advertisement in local paper and internet (via social media), covering the direct surroundings of our clinic (Amsterdam) and by advertisement at the medical faculty of the Academic Medical Center (AMC).

The included subjects will visit the AMC hospital on 3 occasions. During visit 1 the investigators will obtain the Informed consent after oral and written information about the study. The investigators will obtain a medical history, vital signs and laboratory measurements.

During visit 2 the investigators will measure body weight and the investigators will perform an energy expenditure measurement after 40 minutes of bed rest. The investigators will regularly measure temperature by a tympanic thermometer. The subjects will receive intravenous administration of the radioactive pharmacon 18F-FDG, 60 minutes after the administration of the 18F-FDG, and 18F-FDG PET-CT scan will be performed. After the 18F-FDG PET CT scans, the investigators will measure insulin sensitivity by performing an oral glucose tolerance test.

After this visit, subjects will start using bromocriptine (1,25mg/day during the first week and 2,50mg/day during the second week) in the evening.

Visit 3(2 weeks after visit 2) will be exactly the same as visit 2. In the three days before visit 2 and 3, subjects will record their eating behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Caucasian origin
* Subjects should be able and willing to give informed consent
* 18-30 years old
* BMI range of 19-25 kg/m2

Exclusion Criteria:

* Renal failure (creatinine>135mmol/l)
* Liver failure (AST/ (Alanine Aminotransferase) ALT > 3 times higher than the normal upper value)
* Daily use of prescription medication
* Known hypersensitivity to bromocriptine, domperidone maleate or other ergot alkaloids.
* Uncontrolled hypertension
* Known history of coronary artery disease, or other severe cardiovascular conditions (such as a prolonged Qtc-time), or symptoms / history of severe psychiatric disorders.
* Known cardiac valvulopathy
* Prolactin-releasing pituitary tumor (prolactinoma).
* Cases where stimulation of the gastric motility could be harmful: gastro-intestinal haemorrhage, mechanical obstruction or perforation.
* Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not take this medicine.
* Prior participation in a research protocol involving radiation exposure in the last 2 years

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Difference in 18F-FDG uptake before and after using bromocriptin | 17 months
  BAT activity is assessed with a FDG-PET CT scan

SECONDARY OUTCOMES:
Difference in energy expenditure before and after using bromocriptin | 17 months
  energy expenditure is a measure for BAT activity
Difference in core body temperature before and after using bromocriptin | 17 months
  Body temperature might be influenced by BAT activity
Difference in insulin sensitivity before and after using bromocriptin | 17 months
  Insulin sensitivity might be influenced by BAT activity

CONTACTS AND LOCATIONS:
Overall Officials: Frits Holleman, Dr. MD., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands